CLINICAL TRIAL: NCT00472108
Title: A Multicenter, Phase III, Double Blind Study of Photodynamic Therapy (PDT) With Metvix 160 mg/g Cream in Comparison to PDT With Placebo Cream in Patients With Primary Nodular Basal Cell Carcinoma
Brief Title: Photodynamic Therapy (PDT) With Metvix Cream 160 mg/g Versus PDT With Placebo Cream in Participants With Primary Nodular Basal Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PC T307/00; NCT00022503 (obsolete NCT alias)
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Results first posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-02

CONDITIONS: Basal Cell Carcinoma
Keywords: Nodular Basal Cell Carcinoma; Basal Cell Carcinoma; PDT with Metvix 160 mg/g cream; PDT with placebo cream; Histological verification
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Photodynamic Therapy (PDT) WIth Metvix Cream 160 milligrams/gram (mg/g) (Experimental): Participants with BCC lesions were administered to PDT with Metvix® cream 160 mg/g applied topically for three hours, followed by illumination using noncoherent light with a fluency of 75 Joule per centimeter square (J/cm*2) and fluency rate of less than 50-200 milliwatt per centimeter square (mW/cm*2) up to 14 weeks. All participants received two consecutive treatments, one week apart thereby completing one PDT treatment cycle.
  Interventions: Radiation: Photodynamic Therapy (PDT); Drug: Metvix cream
- Placebo Cream (Placebo Comparator): Participants with BCC lesions were administered to PDT with Placebo cream applied topically for three hours, followed by illumination using noncoherent light with a fluency of 75 J/cm*2 and fluency rate of 50-200 mW/cm*2 up to 14 weeks. All participants received two consecutive treatments, one week apart thereby completing one PDT treatment cycle.
  Interventions: Radiation: Photodynamic Therapy (PDT); Drug: Placebo Cream

INTERVENTIONS:
Radiation: Photodynamic Therapy (PDT)
Drug: Metvix cream
  Arms: Photodynamic Therapy (PDT) WIth Metvix Cream 160 milligrams/gram (mg/g)
Drug: Placebo Cream
  Arms: Placebo Cream

SUMMARY:
Photodynamic therapy (PDT) was the selective destruction of abnormal cells through light activation of a photosensitiser in the presence of oxygen. These cells accumulated more photosensitiser than normal cells. The photosensitiser generated reactive oxygen species upon illumination.

For skin diseases, there had been an increasing interest in using precursors of the endogenous photosensitiser protoporphyrin IX (PpIX). The most commonly used precursors have been 5-aminolevulinic acid (ALA) and its derivatives. The present test drug, Metvix, contained the methyl ester of ALA, which penetrated the lesions well and shows high lesion selectivity.

In vitro studies of animal and human tissues had shown significant intracellular formation of photoactive porphyrins after addition of Metvix. The increased photoactive porphyrins levels induced cytotoxic effects in tumour cells after photoactivation.

The primary objective was to compare PDT with Metvix cream to PDT with placebo cream in terms of participants complete response rates based on histologically verified disappearance of the lesions at 6 months after last treatment cycle. Secondary objectives was to compare the two treatments in terms of histological and clinical mean participant response weighted by the number of lesions within a participant, lesion response rates across participants, clinical complete participant response, cosmetic outcome and adverse events.

DETAILED DESCRIPTION:
A participants were randomised to PDT with Metvix cream or PDT with placebo cream. All eligible basal cell carcinoma (BCC) lesions within a participant received same treatment. All participants received two consecutive treatments one week apart. At the 3-months follow-up visit, lesions with no clinical response or progression were surgically excised. Lesions with partial response 50 percent (%) or greater reduction on lesion area) were re-treated; if they do not show complete response three months later, they were surgically excised. Lesions with complete response were surgically excised 6 months after the first or second PDT cycle. All excised tissue specimens were histologically examined.

ELIGIBILITY:
Inclusion Criteria:

A participant with primary, nodular BCC lesion(s) suitable for entry is defined as a participant with

* Clinically diagnosed primary nodular BCC lesion(s).
* Histologically confirmed diagnosis of BCC.
* BCC lesions suitable for simple excision surgery.
* Males or females above 18 years of age.
* Written informed consent.

Exclusion Criteria:

A participant that is ineligible for inclusion is a participant fulfilling any of the following criteria:

* Participants with porphyria.
* Participants with Gorlin's syndrome.
* Participants with Xeroderma pigmentosum.
* Participants concurrently receiving immunosuppressive medication.
* Participants with a history of arsenic exposure.
* Participants with BCC arising in a previous radiated area.
* Known allergy to Metvix, a similar PDT compound or excipients of the cream.
* Participation in other clinical studies either concurrently or within the last 30 days.
* Pregnant or breast-feeding: All women of child-bearing potential must use adequate contraception (e.g. barrier methods, oral contraceptives or intrauterine device) during the treatment period and one month thereafter. In addition, they must have a negative pregnancy test prior to treatment..
* Conditions associated with a risk of poor protocol compliance.

Lesion Exclusion Criteria:

* A nodular BCC lesion in periorbital area, ears and nasolabial fold.
* A nodular BCC lesion with the longest diameter less than 6 millimeter (mm) or larger than 15 mm in face/scalp, larger than 20 mm on extremities and neck and larger than 30 mm on truncus.
* Pigmented nodular BCC lesion(s)
* Morpheaform nodular BCC lesion(s).
* Infiltrating nodular BCC lesion(s).
* Prior treatment of the BCC lesion(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2000-12 (Actual); Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Whitney Tope, MPhil, MD, Principal Investigator — University of Minnesota Hospital and Clinic
Locations (9):
- United States (9):
  - Clinical Research Specialists Inc, Santa Monica, California
  - Department of Dermatology, University of Minnesota Hospital and Clinic, Minneapolis, Minnesota
  - Department of Dermatology, Mayo Medical School, Mayo Clinic, Rochester, Minnesota
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Department of Dermatology, Roswell Park Cancer Institue, Buffalo, New York
  - Northwest Cutaneous Research Specialists, Portland, Oregon
  - DermResearch, Inc., Austin, Texas
  - Texas Dermatology Research Institute, Dallas, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of nine centres and one dermatopathology laboratory in United States were included. Only seven of nine centres enrolled participants.
  Study was conducted from first participant signed informed consent: December 2000 to Last participant last visit: April 2002
Units Other Than Participants: Lesions
Groups:
- Photodynamic Therapy (PDT) With Metvix Cream 160 Milligrams/Gram (mg/g): Participants with basal cell carcinoma (BCC) lesions were administered to PDT with Metvix® cream 160 mg/g applied topically for three hours, followed by illumination using noncoherent light with a fluency of 75 Joule per centimeter square (J/cm*2) and fluency rate of less than 50-200 milliwatt per centimeter square (mW/cm*2) up to 14 weeks. All participants received two consecutive treatments, one week apart thereby completing one PDT treatment cycle.
- Photodynamic Therapy (PDT) With Placebo Cream: Participants with BCC lesions were administered to PDT with Placebo cream applied for three hours, followed by illumination using noncoherent light with a fluency of 75 J/cm*2 and fluency rate of 50-200 mW/cm*2 up to 14 weeks. All participants received two consecutive treatments, one week apart thereby completing one PDT treatment cycle.
Period: Overall Study
Arm/Group | Photodynamic Therapy (PDT) With Metvix Cream 160 Milligrams/Gram (mg/g) | Photodynamic Therapy (PDT) With Placebo Cream
Started | 33; 45 Lesions | 32; 41 Lesions
Completed | 33; 41 Lesions | 31; 39 Lesions
Not Completed | 0; 4 Lesions | 1; 2 Lesions
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Photodynamic Therapy With Metvix Cream 160 Milligrams/Gram (mg/g): Participants with BCC lesions were administered to PDT with Metvix® cream 160 mg/g applied topically for three hours, followed by illumination using noncoherent light with a fluency of 75 J/cm*2 and fluency rate of less than 50-200 mW/cm*2 up to 14 weeks. All participants received two consecutive treatments, one week apart thereby completing one PDT treatment cycle.
- Photodynamic Therapy (PDT) With Placebo Cream: Participants with BCC lesions were administered to PDT with Placebo cream applied topically for three hours, followed by illumination using noncoherent light with a fluency of 75 Joule per centimeter square (J/cm*2) and fluency rate of 50-200 milliwatt per centimeter square (mW/cm*2) up to 14 weeks. All participants received two consecutive treatments, one week apart thereby completing one PDT treatment cycle.
- Total: Total of all reporting groups
Arm/Group | Photodynamic Therapy With Metvix Cream 160 Milligrams/Gram (mg/g) | Photodynamic Therapy (PDT) With Placebo Cream | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Full Range); unit: Years] | 62 [28 to 88] | 67 [39 to 88] | 65 [28 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 25 | 25 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 33 | 32 | 65
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Histologically Confirmed Complete Response
Description: The histological complete response was defined as 100 percent (%) of the lesions within the participant having negative findings in the histological examination. Histological examination included evaluation of all the microscopical slides from the excised tissue for presence of malignant basal cells. Complete response was defined as complete disappearence of lesion. Number of participants with histologically confirmed complete response were reported.
Time Frame: up to 9 months
Population: Intent-to-treat (ITT) population included all participants who had BCC lesions and had received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy (PDT) With Metvix Cream 160 Milligrams/Gram (mg/g) | Photodynamic Therapy (PDT) With Placebo Cream
Number analyzed (Participants) | 33 | 32
Participants | 25 | 11

2. Secondary Outcome: Percentage of Lesions With Histologically Confirmed Complete Lesion Response
Description: Histological response weight means no signs of malignant basal cells in all microscopical slides containing excised tissue. The histologically confirmed complete lesion response were reported.
Time Frame: up to 9 months
Population: ITT population included all participants who had BCC lesions and had received at least one dose of study drug.
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Photodynamic Therapy (PDT) With Metvix Cream 160 Milligrams/Gram (mg/g) | Photodynamic Therapy (PDT) With Placebo Cream
Number analyzed (Participants) | 33 | 32
Number analyzed (Lesions) | 41 | 39
percentage of lesions | 78 | 33

3. Secondary Outcome: Percentage of Lesions With Clinically Confirmed Complete Lesion Response
Description: Clinically confirmed complete lesion response means no signs of malignant basal cells in all microscopical slides containing excised tissue. The clinically confirmed complete lesion response were reported.
Time Frame: up to 9 months
Population: ITT population included all participants who had BCC lesions and had received at least one dose of study drug.
Measure: Number; unit: percentage of Lesions
Units Other Than Participants: Lesions
Arm/Group | Photodynamic Therapy (PDT) With Metvix Cream 160 Milligrams/Gram (mg/g) | Photodynamic Therapy (PDT) With Placebo Cream
Number analyzed (Participants) | 33 | 32
Number analyzed (Lesions) | 41 | 39
percentage of Lesions | 80 | 51

4. Secondary Outcome: Histological Verified Lesions With Complete Response
Description: Histological confirmed complete lesion response means no signs of malignant basal cells in all microscopical slides containing excised tissue. Number of histologically confirmed lesions with complete response were reported.
Time Frame: up to 9 months
Population: ITT population set included all participants who had BCC lesions and received at least one dose of study drug.
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Groups:
- Photodynamic Therapy (PDT) Metvix Cream 160 Milligram/Gram (mg/g): Photodynamic Therapy (PDT) With Metvix Cream 160 (milligram/gram): Participants with basal cell carcinoma (BCC) lesions were administered to photodynamic therapy (PDT) with Metvix® cream 160 milligrams per gram (mg/g) applied for three hours, followed by illumination using noncoherent light with a fluency of 75 Joule per centimeter square (J/cm*2) and fluency rate of less than 50-200 milliwatt per centimeter square (mW/cm*2) up to 14 weeks. All participants received two consecutive treatments, one week apart thereby completing one PDT treatment cycle.
- Photodynamic Therapy (PDT) Placebo Cream: Photodynamic Therapy (PDT) With Placebo Cream: Participants with basal cell carcinoma (BCC) lesions were administered to PDT with Placebo cream applied for three hours, followed by illumination using noncoherent light with a fluency of 75 Joule per centimeter square (J/cm*2) and fluency rate of 50-200 milliwatt per centimeter square (mW/cm*2) up to 14 weeks. All participants received two consecutive treatments, one week apart thereby completing one PDT treatment cycle.
Arm/Group | Photodynamic Therapy (PDT) Metvix Cream 160 Milligram/Gram (mg/g) | Photodynamic Therapy (PDT) Placebo Cream
Number analyzed (Participants) | 33 | 32
Number analyzed (Lesions) | 41 | 39
Lesions | 32 | 13

5. Secondary Outcome: Clinically Verified Lesions With Complete Response
Description: Clinically confirmed complete lesion response means no signs of malignant basal cells in all microscopical slides containing excised tissue. Number of clinically confirmed lesions with complete response were reported.
Time Frame: up to 9 months
Population: ITT population set included all participants who had BCC lesions and received at least one dose of study drug.
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Groups:
- Photodynamic Therapy (PDT) Metvix Cream 160 Milligram/Gram (mg/g): Photodynamic Therapy (PDT) With Metvix Cream 160 (milligram/gram): Participants with BCC lesions were administered to PDT with Metvix® cream 160 mg/g applied for three hours, followed by illumination using noncoherent light with a fluency of 75 J/cm*2 and fluency rate of less than 50-200 mW/cm*2 up to 14 weeks. All participants received two consecutive treatments, one week apart thereby completing one PDT treatment cycle.
- Photodynamic Therapy (PDT) Placebo Cream: Photodynamic Therapy (PDT) With Placebo Cream: Participants with BCC lesions were administered to PDT with Placebo cream applied for three hours, followed by illumination using noncoherent light with a fluency of 75 J/cm*2 and fluency rate of 50-200 mW/cm*2 up to 14 weeks. All participants received two consecutive treatments, one week apart thereby completing one PDT treatment cycle.
Arm/Group | Photodynamic Therapy (PDT) Metvix Cream 160 Milligram/Gram (mg/g) | Photodynamic Therapy (PDT) Placebo Cream
Number analyzed (Participants) | 33 | 32
Number analyzed (Lesions) | 41 | 39
Lesions | 28 | 0

6. Secondary Outcome: Number of Participants With Clinically Evaluated Complete Response
Description: The on-site investigator evaluated the lesion response by comparing to the lesion size before and after treatment. Complete response here means complete disappearance of a lesion. Number of participants for whom one or more lesions had a complete response were reported.
Time Frame: up to 9 months
Population: ITT population set included all participants who had BCC lesions and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy (PDT) With Metvix Cream 160 Milligrams/Gram (mg/g) | Photodynamic Therapy (PDT) With Placebo Cream
Number analyzed (Participants) | 33 | 32
Participants | 28 | 15

7. Secondary Outcome: Number of Participants With Cosmetic Outcome Assessed by Investigator and Participants
Description: Cosmetic outcomes were assessed with regards to occurrence of the following signs or symptoms; scarring, atrophy, induration, redness or change in pigmentation. Cosmetic outcome were graded as excellent, good, fair or poor where: excellent: no scarring, atrophy or induration, no or slight occurrence of redness or change in pigmentation compared to adjacent skin; good: no scarring, atrophy or induration but moderate redness or change in pigmentation compared to adjacent skin; fair: slight to moderate occurrence of scarring, atrophy or induration and Poor: extensive occurrence of scarring, atrophy or induration. The investigator and participants assessed the cosmetic outcome for each lesion has responded completely. Participants were asked to evaluate evaluate the cosmetic outcome according to the same categories: excellent, good, fair cosmetic outcome. Number of participants with summarized cosmetic outcomes for all symptoms as assessed by Investigator and participants were reported.
Time Frame: up to 9 months
Population: ITT population set included all participants who had BCC lesions and received at least one dose of study drug. Here, "Overall Number of participants analyzed" signifies those participants who were evaluable for this outcome measure. Number analyzed = participantswith available data for specified category.
Measure: Count of Participants; unit: Participants
Groups:
- Photodynamic Therapy (PDT) With Metvix Cream 160 Milligram/Gram (mg/g): Participants with basal cell carcinoma (BCC) lesions were administered to PDT with Metvix® cream 160 mg/g applied topically for three hours, followed by illumination using noncoherent light with a fluency of 75 Joule per centimeter square (J/cm*2) and fluency rate of less than 50-200 milliwatt per centimeter square (mW/cm*2) up to 14 weeks. All participants received two consecutive treatments, one week apart thereby completing one PDT treatment cycle.
Arm/Group | Photodynamic Therapy (PDT) With Metvix Cream 160 Milligram/Gram (mg/g) | Photodynamic Therapy (PDT) With Placebo Cream
Number analyzed (Participants) | 28 | 10
Participants
  Excellent: Investigator: number analyzed (Participants) | 28 | 9
  Excellent: Investigator | 17 | 5
  Good: Investigator: number analyzed (Participants) | 28 | 9
  Good: Investigator | 9 | 3
  Fair: Investigator: number analyzed (Participants) | 28 | 9
  Fair: Investigator | 2 | 1
  Poor: Investigator: number analyzed (Participants) | 28 | 9
  Poor: Investigator | 0 | 0
  Excellent: Participant | 18 | 8
  Good: Participant | 8 | 2
  Fair: Participant | 2 | 0
  Poor: Participant | 0 | 0

8. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events (AEs)
Description: Adverse event (AE) was defined as any untoward medical occurrence in a participant, which does not necessarily have causal relationship with treatment. A serious AE was defined as an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged in participant hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs: events between first dose of study drug that were absent before treatment/that worsened relative to pre-treatment state. TEAEs included both serious TEAEs and non-serious TEAEs. Number of participants with AEs and serious AEs were reported.
Time Frame: up to 6 months
Population: The Safety population included all participants in the ITT who were administered at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Photodynamic Therapy (PDT) With Metvix Cream 160 Milligrams/Gram (mg/g) | Photodynamic Therapy (PDT) WIth Placebo Cream
Number analyzed (Participants) | 33 | 32
Participants
  Participants With Adverse Events (AEs) | 30 | 24
  Participants With Serious Adverse Events (AEs) | 1 | 5

ADVERSE EVENTS:
Time Frame: up to 6 months
Description: The Safety population included all participants in the ITT who were administered at least 1 dose of study drug.
Arm/Group | Photodynamic Therapy (PDT) With Metvix Cream 160 Milligrams/Gram (mg/g) | Photodynamic Therapy (PDT) With Placebo Cream
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/33 | 5/32
Other Adverse Events (participants affected / at risk) | 0/33 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Photodynamic Therapy (PDT) With Metvix Cream 160 Milligrams/Gram (mg/g) (N=33) | Photodynamic Therapy (PDT) With Placebo Cream (N=32)
Carotsid Stenosis (Vascular disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Superficial femoral artery to dorsalis (Surgical and medical procedures) | 0 | 1
Redden Ulcer and Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Abdominal aneuryse - ruptured (Gastrointestinal disorders) | 0 | 1
New malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes